CLINICAL TRIAL: NCT02235857
Title: Treatment of Drug-resistant Pediatric Primary Focal Segmental Glomerulosclerosis Using the Liposorber® LA-15 System
Brief Title: Post Approval Study of Liposorber LA-15 System for the Treatment of Focal Segmental Glomerulosclerosis in Children
Acronym: FSGS pediatric
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaneka Medical America LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMA-FSGS-H120005
Record Dates: First submitted 2014-09-06; First posted 2014-09-10 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2024-10

CONDITIONS: Focal Segmental Glomerulosclerosis
Keywords: pediatric, renal transplantation, recurrence, drug-resistant
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Recurrence

STUDY DESIGN:
Intervention Model Description: Patients with focal segmental glomerulosclerosis treated by LIPOSORBER® LA-15 system
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Liposorber® LA-15 System (Experimental): All study patients who meet the study eligibility criteria will undergo the extracorporeal treatment using Liposorber® LA-15 System. The participants are to be treated with the system twice weekly for the 3weeks and then once weekly for the following 6 weeks.
  Interventions: Device: LIPOSORBER® LA-15 System

INTERVENTIONS:
Device: LIPOSORBER® LA-15 System — LIPOSORBER® LA-15 System is an extracorporeal blood purification system. Approximately 3 to 4 L of plasma is treated in a single treatment session and it takes 2 to 3 hours. Recommended frequency of the treatment is twice weekly for 3 weeks followed by once weekly for 6 weeks, thus it takes 9 weeks for a total of 12 treatment sessions.
  Other Names: LDL apheresis; LDL adsorption; dextran sulfate column

SUMMARY:
Liposorber® LA-15 System is a blood purification therapy that selectively removes malignant lipoproteins including low density lipoprotein from circulating blood flow and rapidly reduces the plasma cholesterol level. The system was originally developed for the treatment of patients with serious dyslipidemia such as familial hypercholesterolemia and then applied to improve the dyslipidemia, a common complication of nephrotic syndrome and found to bring about improvement not only with the dyslipidemic condition but the nephrotic condition (e.g, proteinuria and hypoproteinemia).

Although the definitive mechanism by which the system may relieve nephrotic syndrome is unknown, it has been recognized as one of alternative therapies for refractory nephrotic syndrome including focal segmental glomerulosclerosis (FSGS) in Japan and referred in the Guidelines for the Treatment of Nephrotic Syndrome endorsed by The Japanese Society of Nephrology.

This study is conducted as a post approval study imposed by Humanitarian Device Exemption (HDE) order to confirm the safety and efficacy of the Liposorber® LA-15 System in the treatment of drug-resistant pediatric primary FSGS.

ELIGIBILITY:
Inclusion Criteria:

* A pediatric patient is deemed suitable for inclusion in the study if the patient has FSGS with a GFR ≥ 45 ml/min/1.73 m 2 and any of the following:

  * Refractory nephrotic syndrome in which standard treatment options are unsuccessful (i.e., patient is unresponsive to standard corticosteroid and/or calcineurin inhibitor therapy for at least 8 weeks resulting in failure to achieve complete or partial remission);
  * Refractory nephrotic syndrome in which standard treatment options are not well tolerated (i.e., patients intolerant to standard therapies due to severe side effects that negatively affect quality of life without providing an acceptable level of clinical benefit);
  * Refractory or recurrent nephrotic syndrome in which standard therapy is contraindicated.

or

- Pediatric post renal transplant patients with nephrotic syndrome associated with primary FSGS.

Exclusion Criteria:

* General Exclusion Criteria

  * Patient is greater than 21 years of age
  * Parent or patient is unwilling or unable to sign and date the informed consent (Note: Only patients 18-21 years of age may sign the informed consent on their own behalf)
  * Pregnant, lactating, or planning to become pregnant prior to completing the study (Note: The safety of the use of Liposorber® in pregnant women has not been studied. There may be unknown risks to an embryo/fetus. Sexually active women of child bearing potential should avoid pregnancy during the use of the Liposorber device and throughout the study duration.)
  * Unable or unwilling to comply with the follow-up schedule
  * Simultaneously participating in another investigational drug or device study
  * Body weight < 15 kg (33.1 lbs)
* Medical Exclusion Criteria

  * Currently being administered ACE inhibitors that cannot be withheld for at least 24 hours prior to each apheresis treatment (Note: The time period to withhold ACE inhibitors should be prolonged, if determined by the treating physician, considering each individual's renal function and the biological half-life of the ACE-inhibitor currently in use.)
  * Currently being administered antihypertensive drugs other than ACE inhibitors (e.g., Angiotensin II receptor blockers (ARBs) that cannot be withheld on the day of apheresis until after the procedure
  * Medical condition or disorder that would limit life expectancy to less than the primary clinical study endpoint or that may cause noncompliance with the study plan or confound the data analysis
  * Hypersensitivity to dextran sulfate, heparin, or ethylene oxide
  * Adequate anticoagulation cannot be achieved due to severe hemophilia, severe hemorrhage diathesis, severe gastrointestinal ulcers, or are recipients of vitamin K antagonist medications
  * Extracorporeal circulation therapy with Liposorber® LA-15 System cannot be tolerated due to severe cardiac insufficiency, acute myocardial infarction, severe cardiac arrhythmia, acute apoplexy, severe uncontrollable hypertension, or severe uncontrollable hypotension
  * Cardiac impairments such as uncontrolled arrhyth¬mia, unstable angina, decompensated congestive heart failure, or valvular disease
  * Functional thyroid disease or liver abnormalities
  * Unresolved systemic or local infection that could affect the clinical study outcomes

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2015-05-03 (Actual); Primary Completion 2026-05-03 (Estimated); Study Completion 2028-07-03 (Estimated)

PRIMARY OUTCOMES:
The percent of patients who show complete or partial remission | 1 month after the final treatment
the rate of device-related and procedure-related serious adverse events | During the period in which the apheresis procedures are administered and up to at the 1-month follow-up visit

SECONDARY OUTCOMES:
Nephrotic Condition | 1, 3, 6, 12, and 24 months after the final treatment
  Nephrotic condition defined as follows:
  urine protein:creatinine ratio > 2.0 (g/g) with a first morning void urine sample
The percent of patients who obtain complete or partial remission | 3, 6, 12, and 24 months after the final treatment
Incidence of adverse events | From the initiation of the first apheresis session until the termination of the last (usually 12th) apheresis session, standad period of 9 weeks for a total of 12 aoheresis sessions
  The protocol indicates the standard treatment schedule as follows:
  2 sessions weekly for the first 3 weeks followed by 1 session weekly for 6 weeks
Incidence of adverse events and severe adverse events | From 1 months to 24 months after the final aphresis
Various laboratory values | 1,3, 6, 12, and 24 months after the final apheresis
  Various laboratory values include Urine protein, Urine creatinine, Serum creatinine, Estimated glomerular filtration rate (eGFR), serum total protein, Serum albumin, Serum vitamin E, Hematocrit, Red blood cell, White blood cell, Platelet, Total cholesterol, LDL cholesterol, HDL cholesterol, Triglycerides, Serum soluble urokinase plasminogen activator receptor.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey I Silberzweig, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (12):
- United States (12):
  - Loma Linda University Children's Hospital, Loma Linda, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Nemours/A.I. duPont Hospital for Children, Wilmington, Delaware
  - Nemours Children's Health, Orlando, Florida
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Weill Cornell Medical Center / NewYork-Presbyterian, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Medical University of South Carolina Children's Hospital, Charleston, South Carolina
  - Children's Hospital of Richmond at VCU, Richmond, Virginia

REFERENCES:
- [Background] Reidy K, Kaskel FJ. Pathophysiology of focal segmental glomerulosclerosis. Pediatr Nephrol. 2007 Mar;22(3):350-4. doi: 10.1007/s00467-006-0357-2. Epub 2007 Jan 10. PMID 17216262
- [Background] Franceschini N, North KE, Kopp JB, McKenzie L, Winkler C. NPHS2 gene, nephrotic syndrome and focal segmental glomerulosclerosis: a HuGE review. Genet Med. 2006 Feb;8(2):63-75. doi: 10.1097/01.gim.0000200947.09626.1c. PMID 16481888
- [Background] Korbet SM. The treatment of primary focal segmental glomerulosclerosis. Ren Fail. 2000 Nov;22(6):685-96. doi: 10.1081/jdi-100101956. PMID 11104158
- [Background] Tarshish P, Tobin JN, Bernstein J, Edelmann CM Jr. Cyclophosphamide does not benefit patients with focal segmental glomerulosclerosis. A report of the International Study of Kidney Disease in Children. Pediatr Nephrol. 1996 Oct;10(5):590-3. doi: 10.1007/s004670050167. PMID 8897562
- [Background] Fine RN. Recurrence of nephrotic syndrome/focal segmental glomerulosclerosis following renal transplantation in children. Pediatr Nephrol. 2007 Apr;22(4):496-502. doi: 10.1007/s00467-006-0361-6. Epub 2006 Dec 21. PMID 17186280
- [Background] Schwartz GJ, Munoz A, Schneider MF, Mak RH, Kaskel F, Warady BA, Furth SL. New equations to estimate GFR in children with CKD. J Am Soc Nephrol. 2009 Mar;20(3):629-37. doi: 10.1681/ASN.2008030287. Epub 2009 Jan 21. PMID 19158356
- [Background] Trachtman H, Vento S, Gipson D, Wickman L, Gassman J, Joy M, Savin V, Somers M, Pinsk M, Greene T. Novel therapies for resistant focal segmental glomerulosclerosis (FONT) phase II clinical trial: study design. BMC Nephrol. 2011 Feb 10;12:8. doi: 10.1186/1471-2369-12-8. PMID 21310077